CLINICAL TRIAL: NCT04449861
Title: An Open Label, Multicenter Study of First-Line Durvalumab Plus Platinum-Based Chemotherapy in Chinese Patients With Extensive Stage Small-Cell Lung Cancer (Oriental)
Brief Title: Durvalumab Plus Chemotherapy in ES-SCLC (Oriental)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D419BR00018
Record Dates: First submitted 2020-05-06; First posted 2020-06-29 (Actual); Results first posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Small Cell Lung Carcinoma Extensive Disease
MeSH Terms: interventions — durvalumab; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Durvalumab plus 4-6 cycles chemotherapy (Experimental): Participants will receive treatment with durvalumab + etoposide and either cisplatin or carboplatin (EP) for 4 to 6 cycles. Durvalumab will be administered at a dose of 1500 mg every 3 weeks (Q3W) with first-line chemotherapy (EP) and will continue to be administered as monotherapy every 4 weeks (Q4W) post-chemotherapy until progressive disease (PD). Prophylactic cranial irradiation (PCI) is allowed at the investigators' discretion as per SoC guidance for ES-SCLC. Patients will attend a safety follow up visit 90 days after last dose of durvalumab.
  Interventions: Drug: Durvalumab plus chemotherapy

INTERVENTIONS:
Drug: Durvalumab plus chemotherapy — Drug: Durvalumab IV infusions every 3 weeks for 4-6 cycles and every 4 weeks thereafter until PD or other discontinuation criteria.
  Drug: Carboplatin 4-6 cycles every 3 weeks
  Drug: Cisplatin 4-6 cycles every 3 weeks
  Drug: Etoposide 4-6 cycles every 3 weeks

SUMMARY:
This will be an open-label, single-arm, multicenter, Phase IIIb study to determine the safety of durvalumab + etoposide and cisplatin or carboplatin as first-line treatment in patients with extensive stage small-cell lung cancer.

ELIGIBILITY:
For inclusion in the study, patients should fulfill the following criteria:

1. Male or female ≥18 years at the time of Screening.
2. Written informed consent obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.
3. Histologically or cytologically documented extensive stage SCLC (stage IV [T any, N any, M1 a/b], or with T3-4 due to multiple lung nodules that are too extensive or have tumor/nodal volume that is too large to be encompassed in a tolerable radiation plan, according to American Joint Committee on Cancer Stage 8th edition).

   - Brain metastases; must be asymptomatic or treated and stable off steroids and anti-convulsants for at least 1 month prior to study treatment. Patients with suspected brain metastases at screening should have a CT/MRI of the brain prior to study entry.
4. Patients must be considered suitable to receive a platinum-based chemotherapy regimen as 1st line treatment for the ES-SCLC. Chemotherapy must contain either cisplatin or carboplatin in combination with etoposide.
5. Life expectancy ≥12 weeks at Day 1.
6. World Health Organization (WHO)/Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2 at enrollment.

   - Note: Patients with PS2 will be limited to a maximum of 20% of the total study population; once this limit is met, additional enrolled patients must have PS 0-1.
7. Body weight >30 kg.
8. At least 1 lesion, not previously irradiated, that can be accurately measured at baseline as ≥10 mm in the longest diameter (except lymph nodes which must have a short axis ≥15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) and that is suitable for accurate repeated measurements as per RECIST 1.1 guidelines.
9. Baseline CT/MRI results of the chest and abdomen (including liver and adrenal glands) within 28 days prior to the treatment initiation.
10. No prior exposure to immune-mediated therapy including, but not limited to, other anti-CTLA-4, anti-PD-1, anti-PD-L1, and anti-programmed cell death ligand 2 (anti-PD-L2) antibodies, excluding therapeutic anticancer vaccines.
11. Adequate organ and marrow function as defined below (test can be repeated once if necessary):

    * Hemoglobin ≥9.0 g/dL.
    * Absolute neutrophil count ≥1.5 × 10^9/L (use of granulocyte colony-stimulating factor is not permitted at within 7 days before testingscreening).
    * Platelet count ≥100 × 10^9/L.
    * Serum bilirubin ≤1.5 × the upper limit of normal (ULN).
    * In patients without hepatic metastasis: ALT and AST ≤2.5 × ULN.
    * In patients with hepatic metastases, ALT and AST ≤5 × ULN.
    * Measured or calculated creatinine clearance: >60mL/min for patients planned to be treated with cisplatin and >40mL/min for patients planned to be treated with carboplatin
12. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause.

The following age-specific requirements apply:

* Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
* Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).

Patients should not enter the study if any of the following exclusion criteria are fulfilled:

1. Previous IP assignment in the present study.
2. Medical contraindication to etoposide-platinum (carboplatin or cisplatin)-based chemotherapy.
3. Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
4. Received prior systemic therapy for ES-SCLC. Patients who have received prior chemoradiotherapy for limited-stage SCLC must have been treated with curative intent and experienced a treatment-free interval of at least 6 months since last chemotherapy, radiotherapy, or chemoradiotherapy cycle from diagnosis of ES-SCLC
5. Any condition that, in the opinion of the treating physician, would interfere with evaluation of the study drug or interpretation of patient safety.
6. Planned consolidation chest radiation therapy. Radiation therapy outside of the chest for palliative care (ie, bone metastasis) is allowed but must be completed before first dose of the study medication.
7. Major surgical procedure (as defined by the investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.
8. History of allogeneic organ transplantation.
9. Has a paraneoplastic syndrome (PNS) of autoimmune nature, requiring systemic treatment (systemic steroids or immunosuppressive agents) or has a clinical symptomatology suggesting worsening of PNS.
10. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis with the exception of diverticulosis, systemic lupus erythematosus, sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, and uveitis, etc]). The following are exceptions to this criterion:

    * Patients with vitiligo or alopecia
    * Patients with hypothyroidism (eg, following Hashimoto syndrome) and stable on hormone replacement
    * Any chronic skin condition that does not require systemic therapy
    * Patients without active disease in the last 5 years may be included but only after consultation with the Study Physician
    * Patients with celiac disease controlled by diet alone
11. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, uncontrolled cardiac arrhythmia, active interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
12. History of active primary immunodeficiency.
13. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis testing in line with local practice), hepatitis B (known positive HBV surface antigen [HbsAg] result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HbsAg) are eligible. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
14. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

    * Intranasal, inhaled, topical steroids or local steroid injections (eg, intra articular
    * injection).
    * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent.
    * Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication). Premedication with steroids for chemotherapy is acceptable.
15. Receipt of live, attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
16. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from Screening to 90 days after the last dose of durvalumab.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (27):
- China (27):
  - Research Site, Baoding
  - Research Site, Changchun
  - Research Site, Chengdu
  - Research Site, Dalian
  - Research Site, Dongyang
  - Research Site, Guangdong
  - Research Site, Guangzhou
  - Research Site, Haerbin
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Huai'an
  - Research Site, Jiangyin
  - Research Site, Jinan
  - Research Site, Jinhua
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Ningbo
  - Research Site, Qingdao
  - Research Site, Shanghai
  - Research Site, Shenzhen
  - Research Site, Taizhou
  - Research Site, Tianjin
  - Research Site, Whenzhou
  - Research Site, Wuhan
  - Research Site, Wuxi
  - Research Site, Yangzhou
  - Research Site, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D419BR00018&attachmentIdentifier=bea5d0f0-7872-4ddc-8841-04bef355afc5&fileName=CSR_synophsis_Redacted.pdf&versionIdentifier=
- See also: Redacted Statistical Analysis Plan — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D419BR00018&attachmentIdentifier=8aab5cc6-2724-45a4-b01d-d43437179031&fileName=Statistical_Analysis_Plan,_ANGEL.pdf&versionIdentifier=
- See also: Redacted Clinical Study Protocol — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D419BR00018&attachmentIdentifier=865699ee-8b5c-414d-8ad6-f245f3ac2534&fileName=SCLC_treatment_study_China_CSP_v2.0_EN_clean_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study recruited the first participant on 07 December 2020 and the last participant's last visit was completed on 30 March 2023. A total of 193 participants were screened, among which, 166 participants (86.0%) were successfully enrolled into the study from 32 study sites in China
Pre-assignment Details: Among the 166 enrolled participants, 165 of them (99.4%) received the study treatment, while only 1 participant (0.6%) did not receive the study treatment.
  All subjects who received at least 1 dose of study treatment will be included in the safety analysis set, which will be the primary analysis set for all analyses.
Groups:
- Durvalumab With EP: durvalumab + etoposide and cisplatin or carboplatin
Period: Overall Study
Arm/Group | Durvalumab With EP
Started (07 December 2020) | 166
Completed (30 March 2023) | 45 (45 participants still in the study when study complete)
Not Completed | 121
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 5
Not completed — Death | 112

BASELINE CHARACTERISTICS:
Population: 165 participants who received at least 1 dose of study treatment were included in baseline analysis population
Arm/Group | Durvalumab With EP
Number analyzed (Participants) | 165
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age (years) | 63.70 (7.699)
Sex: Female, Male [Count of Participants; unit: Participants]
  Sex: Female | 25
  Sex: Male | 140
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 165
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 165
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Grade ≥3 AEs
Time Frame: 19 months
Population: 165 subjects who received at least 1 dose of study treatment are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Durvalumab With EP
Number analyzed (Participants) | 165
percentage of participants | 49.7

2. Primary Outcome: Percentage of Participants With Immune-mediated Adverse Events (imAEs)
Description: An immune-mediated adverse event (imAE) is defined as an AESI that is associated with drug exposure and is consistent with an immune-mediated mechanism of action and where there is no clear alternate aetiology.
Time Frame: 19 months
Population: 165 subjects who received at least 1 dose of study treatment are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Durvalumab With EP
Number analyzed (Participants) | 165
percentage of participants | 24.2

3. Secondary Outcome: Median Progression Free Survival (PFS)
Description: PFS by investigator assessment according to RECIST v1.1 criteria
  Progression-free survival is defined as the time from first dose of study treatment until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the patient withdraws from study therapy or receives another anti-cancer therapy prior to progression. Patients who have not progressed or died at the time of analysis will be censored at the time of the latest date of assessment of investigator. However, if the patient progresses or dies after 2 or more missed visits, the patient will be censored at the time of the latest assessment. If the patient has no evaluable visits or does not have baseline data, they will be censored at the day of first dose unless they die within 2 visits of baseline.
Time Frame: 19 months
Population: 165 subjects who received at least 1 dose of study treatment are included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab With EP
Number analyzed (Participants) | 165
months | 6.3 [5.6 to 6.5]

4. Secondary Outcome: Proportion of Patients Alive and Progression Free at 12 Months (APF12)
Description: The APF12 is defined as the Kaplan-Meier estimate of PFS (per investigator assessment according to RECIST v1.1 criteria) at 12 months.
Time Frame: 12 months
Population: 165 subjects who received at least 1 dose of study treatment are included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Durvalumab With EP
Number analyzed (Participants) | 165
percentage of participants | 17.6 [12.0 to 24.1]

5. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective Response Rate is defined as the number (%) of patients with measurable disease with at least 1 visit response of CR or PR. Data obtained up until progression or last evaluable assessment in the absence of progression will be included in the assessment of ORR. Any CR or PR which occurred after a further anti-cancer therapy was received will not be included in the numerator for the ORR calculation.
Time Frame: 19 months
Population: 165 subjects who received at least 1 dose of study treatment are included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Durvalumab With EP
Number analyzed (Participants) | 165
percentage of participants | 76.4 [69.1 to 82.6]

6. Secondary Outcome: Median Overall Survival (OS)
Description: Overall survival is defined as the time from the date of first dose of study treatment until death due to any cause. Any patient not known to have died at the time of analysis will be censored based on the last recorded date on which the patient was known to be alive.
Time Frame: 19 months
Population: 165 subjects who received at least 1 dose of study treatment are included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab With EP
Number analyzed (Participants) | 165
months | 14.8 [13.2 to 16.0]

7. Secondary Outcome: Proportion of Patients Alive at 12 Months (OS12)
Description: The OS12 is defined as the Kaplan-Meier estimate of OS at 12 months
Time Frame: 12 months
Population: 165 subjects who received at least 1 dose of study treatment are included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Durvalumab With EP
Number analyzed (Participants) | 165
percentage of participants | 60.8 [52.8 to 67.9]

8. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response is defined as the time from the date of first documented response until the date of documented progression or death in the absence of disease progression. The end of response should coincide with the date of progression or death from any cause used for the PFS endpoint. The time of the initial response will be defined as the latest of the dates contributing towards the first visit response of PR or CR.
Time Frame: 19 months
Population: Duration of response is only calculated for patients who have a best overall tumor response of CR or PR before further anti-cancer therapy after first dose.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Durvalumab With EP (CR+PR): Patients who have a best overall tumor response of CR or PR before further anti-cancer therapy after first dose.
Arm/Group | Durvalumab With EP (CR+PR)
Number analyzed (Participants) | 126
months | 5.1 [4.7 to 5.7]

9. Secondary Outcome: Percentage of Participants With AEs
Time Frame: 19 months
Population: 165 subjects who received at least 1 dose of study treatment are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Durvalumab With EP
Number analyzed (Participants) | 165
percentage of participants | 97.6

10. Secondary Outcome: Percentage of Participants With SAEs
Time Frame: 19 months
Population: 165 subjects who received at least 1 dose of study treatment are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Durvalumab With EP
Number analyzed (Participants) | 165
percentage of participants | 42.4

11. Secondary Outcome: Percentage of Participants With Adverse Events of Special Interest (AESI)
Time Frame: 19 months
Population: 165 subjects who received at least 1 dose of study treatment are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Durvalumab With EP
Number analyzed (Participants) | 165
percentage of participants | 40.0

12. Secondary Outcome: Percentage of Participants With AEs Resulting in Treatment Discontinuation
Time Frame: 19 months
Population: 165 subjects who received at least 1 dose of study treatment are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Durvalumab With EP
Number analyzed (Participants) | 165
percentage of participants | 12.1

ADVERSE EVENTS:
Time Frame: 19 months
Arm/Group | Durvalumab With EP
All-Cause Mortality (participants affected / at risk) | 112/165
Serious Adverse Events (participants affected / at risk) | 70/165
Other Adverse Events (participants affected / at risk) | 161/165
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab With EP (N=165)
Anaemia (Blood and lymphatic system disorders) | 15 (16)
Myelosuppression (Blood and lymphatic system disorders) | 8 (8)
Platelet count decreased (Investigations) | 14 (19)
Neutrophil count decreased (Investigations) | 6 (6)
White blood cell count decreased (Investigations) | 6 (7)
Pneumonia (Infections and infestations) | 7 (7)
Urinary tract infection (Infections and infestations) | 2 (3)
Cerebral infarction (Nervous system disorders) | 2 (2)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Agranulocytosis (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Death (General disorders) | 3 (3)
Pyrexia (General disorders) | 2 (2)
Oedema peripheral (General disorders) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Febrile infection (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Hepatitis E (Infections and infestations) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1)
Immune-mediated encephalitis (Nervous system disorders) | 1 (1)
Lacunar infarction (Nervous system disorders) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Immune-mediated hepatic disorder (Hepatobiliary disorders) | 1 (1)
Liver injury (Hepatobiliary disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Aortic dissection (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 1 (1)
Superior vena cava occlusion (Vascular disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Immune-mediated endocrinopathy (Endocrine disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Immune-mediated nephritis (Renal and urinary disorders) | 1 (1)
Otolithiasis (Ear and labyrinth disorders) | 1 (1)
Mania (Psychiatric disorders) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab With EP (N=165)
anaemia (Blood and lymphatic system disorders) | 125 (214)
nausea (Gastrointestinal disorders) | 45 (77)
vomiting (Gastrointestinal disorders) | 36 (64)
alopecia (Skin and subcutaneous tissue disorders) | 36 (36)
constipation (Gastrointestinal disorders) | 35 (49)
decreased appetite (Metabolism and nutrition disorders) | 34 (51)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-03-31): https://cdn.clinicaltrials.gov/large-docs/61/NCT04449861/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-06): https://cdn.clinicaltrials.gov/large-docs/61/NCT04449861/SAP_001.pdf